CLINICAL TRIAL: NCT03690401
Title: Assessment of Body Composition in Cancer Patients Post-Treatment Using the SOZO Device
Brief Title: Body Composition Post Cancer Treatment
Acronym: PostSOZO
Status: Completed | Type: Observational
Sponsor: Prisma Health-Upstate (Other)
Collaborators: ImpediMed Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00077373
Record Dates: First submitted 2018-08-10; First posted 2018-10-01 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Cancer
Keywords: Cancer; Post-Treatment; Body Composition; SOZO; Impedimed
MeSH Terms: conditions — Neoplasms | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Moving On Group: Participants' body composition will be estimated using a SOZO device at 5 different time points over 12 weeks. Participant will also complete questionnaires and physical assessments during each study visit. These include waist & hip measurements, weight/BMI, brief fatigue inventory, timed up and go test, 6 minute walk test, cancer distress assessment, ECOG performance status, hand grip strength test, and 3-day food diary. DEXA scans will be performed before treatment and after completion of treatment. Moving On assessments will be performed at first and last study visits.
  Interventions: Device: SOZO Device; Device: DEXA Scan
- Non-Moving On Group: Participants' body composition will be estimated using a SOZO device at 5 different time points over 12 weeks. Participant will also complete questionnaires and physical assessments during each study visit. These include waist & hip measurements, weight/BMI, brief fatigue inventory, timed up and go test, 6 minute walk test, cancer distress assessment, ECOG performance status, hand grip strength test, and 3-day food diary. DEXA scans will be performed at first and last study visits.
  Interventions: Device: SOZO Device; Device: DEXA Scan

INTERVENTIONS:
Device: SOZO Device — SOZO device will estimate fluid status, total body composition, metabolic report, skeletal muscle mass, phase angle, body mass index, weight, and hydration index analysis. Participants will be asked to fast for at least 8 hours before each visit, but water may be consumed to ensure they are well-hydrated. Participants will be asked to provide a urine sample at each visit and to report the color of your urine to the staff so they can determine how well hydrated the participants are. If not hydrated to the extent needed, participants will be asked to drink water and repeat the urine sample again after 30 minutes. A total of 5 SOZO measurements will be recorded over 12 weeks.
Device: DEXA Scan — DEXA scan bone density reading with hip and spine measurements as well as a whole body composition scan will be performed. Where DEXA cannot be collected on the same day as other study assessments, Weight/BMI, Urine Color, and SOZO should all be collected (or repeated if already done) to coincide with the DEXA scan if SOZO is available at DEXA location.

SUMMARY:
The purpose of this study is to assess how bone density and body composition changes after a cancer patient completes treatment and through 12-weeks post-treatment. Patients who enroll in the 12-week exercise program, Moving On, and those that do not elect to participate in the Moving On program will both be tracked, with assessments including SOZO measurements, DEXA scan (bone density and whole body composition), performance status tests, food log, urine color test, and other study assessments.

DETAILED DESCRIPTION:
This is an observational, prospective, parallel-arm device use study. 50 subjects will be enrolled in the study. The study will look at the changes in the participants body composition post cancer treatment using the SOZO device. The SOZO device is intended to estimate the following body composition parameters: Fluid status (TBW, ECF, ICF), Total body composition (fat free mass, fat mass, % of weight), Metabolic report (active tissue mass, extracellular mass, basal metabolic rate), Skeletal muscle mass, Phase angle, Body mass index (BMI), Weight, and Hydration index (Hy-Dex) analysis. Participants will have 5 study visits during 12 weeks where SOZO measurements will be taken as well as other study measurements.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to provide consent
* Mentally and physically able to comply with protocol
* Age 18 and over
* Body Mass Index (BMI) ≤ 40 or body weight of <300 pounds
* Recent diagnosis of first cancer stage I-III
* Completion of final primary cancer treatment within 6 months of Screening/Baseline visit

Exclusion Criteria:

* Active implanted medical device (cardiac pacemakers, defibrillators) or connected to electronic life support devices or patients with other metallic devices that would interfere with BIS measurements
* Amputees
* Any acute swelling condition diagnosed or actively being treated within 30 days of screening/baseline (including, but not limited to: acute heart failure, renal disease with dialysis, pulmonary edema, thrombophlebitis, deep vein thrombosis, pleural effusion, ascites, pregnancy)
* Patients with basal cell carcinoma or squamous cell skin cancer
* Patients with head or neck cancer
* Currently suffering from uncontrolled intercurrent illness, including: ongoing/active infection, unstable angina pectoris, or cardiac arrhythmia
* Enrollment of female breast cancer patients not to exceed 60% of total projected enrollment. Once this threshold has been reached, these subjects will be excluded
* Planned orthopedic implant surgery
* Planned breast implant surgery
* Presence of or plan for breast expanders post-mastectomy
* Dependent upon transfusions
* Any history of organ transplant
* Presence of colostomy/ostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients who received their first diagnosis of most cancer types stage I-III. Patients must have recently completed their cancer treatment and be eligible to participate in the Moving On program, although patient will be eligible to participation in this study regardless of willingness to participate in the Moving On program. Non-Moving On program participants must constitute ≥ 10 and ≤ 25 of the overall enrolled patient population to ensure adequate controls are in place.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
SOZO device can detect changes in body composition using SOZO measurements. | 12 weeks
  Change from baseline in body composition measures (intracellular fluid, extracellular fluid, fat mass, fat free mass, skeletal muscle mass, phase angle, and hydration index)

SECONDARY OUTCOMES:
Patient general health | 12 weeks
  Evaluate patient general health using physical performance tests
Correlate SOZO with food recall. | 12 weeks
  Assess correlation of SOZO measurements with 3-day food recall.
Correlate SOZO with DEXA Scan | 12 weeks
  Assess correlation of SOZO measurements and DEXA scan (bone density with hip and spine measurements and whole body composition) results.
Correlate SOZO with standard of care | 12 weeks
  Assess correlation of SOZO measurements with standard of care measurements.
Detect changes in participant fatigue | 12 weeks
  Change from baseline in Brief Fatigue Inventory score
Detect changes in participant stress | 12 weeks
  Change from baseline in Suscro Distress Inventory score
Correlate SOZO with urine test. | 12 weeks
  Assess correlation of SOZO measurements with urine color test.

CONTACTS AND LOCATIONS:
Overall Officials: Larry Gluck, MD, Principal Investigator — Prisma Health
Locations (1):
- Prisma Health Cancer Institute Center for Integrative Oncology and Survivorship, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mayer DK, Nasso SF, Earp JA. Defining cancer survivors, their needs, and perspectives on survivorship health care in the USA. Lancet Oncol. 2017 Jan;18(1):e11-e18. doi: 10.1016/S1470-2045(16)30573-3. PMID 28049573
- [Background] Jacobs LA, Shulman LN. Follow-up care of cancer survivors: challenges and solutions. Lancet Oncol. 2017 Jan;18(1):e19-e29. doi: 10.1016/S1470-2045(16)30386-2. PMID 28049574